CLINICAL TRIAL: NCT05540860
Title: A 2-part Phase 2 Study of Safety, Pharmacokinetics and Biomarkers in Children With Duchenne Muscular Dystrophy Including a Randomized, Double-Blind, Placebo-Controlled Part A, Followed by an Open-Label Part B
Brief Title: A Study of EDG-5506 in Children With Duchenne Muscular Dystrophy (LYNX)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDG-5506-210
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 1; Drug: Placebo
- Cohort 2 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 2; Drug: Placebo
- Cohort 3 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 3; Drug: Placebo
- Cohort 4 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 4; Drug: Placebo
- Cohort 5 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 5; Drug: Placebo
- Cohort 2NS (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 2; Drug: Placebo

INTERVENTIONS:
Drug: Sevasemten Dose 1 — Sevasemten is administered orally once per day
  Arms: Cohort 1
Drug: Sevasemten Dose 2 — Sevasemten is administered orally once per day
  Arms: Cohort 2; Cohort 2NS
Drug: Sevasemten Dose 3 — Sevasemten is administered orally once per day
  Arms: Cohort 3
Drug: Sevasemten Dose 4 — Sevasemten is administered orally once per day
  Arms: Cohort 4
Drug: Sevasemten Dose 5 — Sevasemten is administered orally once per day
  Arms: Cohort 5
Drug: Placebo — Placebo is administered orally once per day

SUMMARY:
The LYNX study is a 2-part, multicenter, Phase 2 study of safety, pharmacokinetics and biomarkers in children with Duchenne muscular dystrophy including a randomized, double-blind, placebo-controlled part A, followed by an open-label part B.

DETAILED DESCRIPTION:
This is a 2-part, multi-center, Phase 2 study to evaluate the effect of sevasemten (EDG-5506) on safety, pharmacokinetics and biomarkers of muscle damage in approximately 72 children with DMD treated with oral, once-daily sevasemten for up to 48 months. This study will have up to a 4-week Screening period, a 12-week randomized, double-blind, placebo controlled treatment period (Part A), up to a 196-week open-label extension period (Part B), and a 2-week follow up period.

Approximately 72 participants aged 4 to 9 years inclusive will be randomized to sevasemten or placebo in a 2:1 ratio. Five dose cohorts (C1, C2, C3, C4 and C5) of approximately 9 participants each will be enrolled sequentially. Approximately 18 total additional participants may be added across Cohorts 2, 3, or 4.

An additional cohort, Cohort 2NS, to include participants (aged 4 to 7 years inclusive) not currently treated with corticosteroids, will enroll approximately 9 participants after Cohort 2 safety review and in parallel with the additional cohorts.

After review of emerging data, the protocol was amended so all dose cohorts receive the same dose in Part B.

ELIGIBILITY:
Key Common Inclusion Criteria:

1. A documented mutation on the DMD gene and phenotype consistent with Duchenne muscular dystrophy.
2. Able to complete the stand from supine in ≤ 10 seconds and able to perform the 4-stair climb in < 10 seconds at the Screening visit.
3. Body weight greater than or equal to 15 kg at the Screening visit.

For Cohorts 1, 2, 3, 4 and 5:

Aged 4-9 years on a stable dose of corticosteroids for a minimum of 6 months prior to the Baseline visit.

For Cohort 2 Non-Steroid (Cohort 2NS):

Aged 4-7 years not on corticosteroids within 6 months prior to the Baseline visit.

Key Common Exclusion Criteria:

1. Medical history or clinically significant physical exam/laboratory result that, in the opinion of the investigator, would render the participant unsuitable for the study. This includes venous access that would be too difficult to facilitate repeated blood testing.
2. A forced vital capacity < 60% predicted at the Screening visit for those participants who are > 8 years old at Screening.
3. A cardiac echocardiography showing left ventricular ejection < 45% at the Screening visit.
4. Receipt of an investigational drug within 30 days or 5 half-lives (whichever is longer) of the Screening visit in the present study.
5. Receipt of a stable dose of an approved exon-skipping therapy with a treatment duration of less than 1 year prior to the Screening visit.

For Cohort 2 Non-Steroid (Cohort 2NS):

Receipt of oral corticosteroids for the treatment of Duchenne muscular dystrophy in the previous 6 months. Participants will not be tapered off steroids for the purpose of this study and oral corticosteroids for the treatment of Duchenne muscular dystrophy may be initiated after the Week 16 visit.

Ages: 4 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events during treatment with sevasemten or placebo | 48 months
  All participants
Severity of adverse events during treatment with sevasemten or placebo | 48 months
  All participants

SECONDARY OUTCOMES:
Incidence of laboratory test-related treatment emergent adverse events | 48 months
  All participants
Pharmacokinetics as measured by steady state plasma concentration | 48 months
  All participants
Change from Baseline in serum creatinine kinase | 12 weeks
  All participants
Change from Baseline in fast skeletal muscle troponin I | 12 weeks
  All participants

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://edgewisetx.com